CLINICAL TRIAL: NCT00006324
Title: Hormonal Contraception and the Risk of HIV Acquisition
Brief Title: Hormonal Birth Control and the Risk of Acquiring HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: HIVNET 021
Record Dates: First submitted 2000-10-02; First posted 2001-08-31 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2006-11

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; Delayed-Action Preparations; Risk Factors; Prevalence; Contraceptive Agents, Female; Contraceptives, Oral, Combined; Medroxyprogesterone 17-Acetate
MeSH Terms: conditions — HIV Infections | interventions — Ethinyl Estradiol-Norgestrel Combination; Medroxyprogesterone Acetate

INTERVENTIONS:
Drug: Ethinyl estradiol/levonorgestrel
Drug: Medroxyprogesterone acetate

SUMMARY:
The purpose of this study is to find out whether hormonal birth control increases, decreases, or does not change the risk of women becoming infected with HIV.

Sexual intercourse between men and women is the main way HIV is transmitted. About 90 percent of HIV infections in women are caused by sexual intercourse. Also, hormonal birth controls are widely used. This study hopes to find out whether hormonal birth control changes the risk of women becoming infected with HIV.

DETAILED DESCRIPTION:
Heterosexual intercourse is the primary mode of HIV transmission worldwide and accounts for about 90% of HIV infections in women. Hormonal contraceptives including COCs and injectables are among the most widely used contraceptives in the world. Understanding the impact of hormonal contraception on HIV transmission is a critical unanswered public health question. Because of the critical nature of this issue to women of reproductive age worldwide, a methodologically sound study must be undertaken. It must be determined if hormonal contraceptive use increases the risk of HIV infection and the magnitude of the association, if it exists.

This study takes place in Thailand, Uganda, and Zimbabwe. HIV-seronegative women continue using their current birth control method (low dose COC, DMPA injections, or non-hormonal contraceptive methods [condoms, sterilization, or no modern contraception method]) for the duration of the study. They are followed every 12 weeks for a minimum of 15 months and a maximum of 24 months, or until seroconversion. Pelvic exams, including Pap smears, are done, blood samples are drawn, and vaginal and cervical specimens are tested for any sexually transmitted diseases (STDs). Women are provided with free treatment for any STDs that are diagnosed. They complete a questionnaire on sexual behavior and contraceptive history; counseling on contraceptive use and reducing HIV risk is provided.

ELIGIBILITY:
Inclusion Criteria

Women may be eligible for this study if they:

* Are 16 to 35 years of age.
* Attend family planning and maternal and child health clinics in Zimbabwe, Thailand, or Uganda.
* Have been using low-dose birth control pills, DMPA injections, or non-hormonal birth control (condoms, sterilization, or no modern birth control method) for at least 3 months and plan to continue using the same type of birth control for a year.
* Are HIV-negative.
* Are sexually active.
* Are at least 4.5 months after delivery, if they have given birth.
* Agree to all study procedures, including HIV testing every 3 months, follow-up clinic visits, and home visits if they fail to return for follow-up.
* Have a home address where they can be reached for follow-up visits.

Exclusion Criteria

Women will not be eligible for this study if they:

* Are pregnant or plan to try to become pregnant in the next year. Women who become pregnant after enrolling in the trial will not be discontinued.
* Are not currently using low-dose birth control pills or DMPA for birth control but have used low-dose birth control pills within the last 3 months, or DMPA for birth control within the previous 6 months.
* Are HIV-indeterminate or HIV-positive.
* Have used an IUD for birth control in the last month.
* Have used non-study types of birth control (such as Norplant, NET-EN, or progestin-only pills) within the last 3 months.
* Have had a full hysterectomy.
* Have had an abortion or miscarriage within the last month.
* Have had a blood transfusion within the last 3 months.
* Were previously or are currently in an HIV vaccine trial.
* Injected illegal drugs within the last 3 months.

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6360
Dates: Start 1999-12; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Overall Officials: Charles Morrison, Study Chair; Barbra Richardson, Study Chair; Sungwal Rugpao, Principal Investigator; Roy Mugerwa, Principal Investigator; Francis Mmiro, Principal Investigator; Tsungai Chipato, Principal Investigator
Locations (1):
- Amy Lovvorn, Research Triangle Park, North Carolina, United States